CLINICAL TRIAL: NCT03022747
Title: Optimizing 6-mercaptopurine Therapy in Pediatric Acute Lymphoblastic Leukemia by Using Allopurinol Clinical Study in Children 1-19 Years on Maintenance Therapy for Acute Lymphoblastic Leukemia.
Brief Title: Optimizing 6-mercaptopurine Therapy in Pediatric Acute Lymphoblastic Leukemia by Using Allopurinol
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Allopurinol Study V3.0
Record Dates: First submitted 2017-01-09; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard maintenance therapy (Active Comparator): Standard maintenance therapy with 6 mercaptopurine and methotrexate
  Interventions: Drug: Standard treatment
- Allopurinol treatment (Experimental): The second 12 week phase during which allopurinol is added to oral 6-mercaptopurine and methotrexate therapy
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol is added to standard oral 6-mercaptopurine and methotrexate
  Arms: Allopurinol treatment
Drug: Standard treatment — Oral 6-mercaptopurine and methotrexate
  Arms: Standard maintenance therapy

SUMMARY:
The study will investigate, in children with acute lymphoblastic leukemia during maintenance treatment, if addition of allopurinol to conventional oral 6-mercaptopurine and methotrexate therapy, affects erythrocyte concentrations of 6-thioguanine and 6 methylmercaptopurine. The effect on hematological and liver toxicity parameters in blood will also be investigated as well as clinical toxicity.

DETAILED DESCRIPTION:
After one month of conventional maintenance therapy (MT) children and adolescents, treated for acute lymphoblastic leukemia on Nordic protocols and with wild type thiopurine methyltransferase (TPMT) are eligible for the study. They will first receive a 12 week phase with normal MT during which time repeated sampling of 6-mercaptopurine (6MP) metabolite levels and other laboratory parameters will be performed. After 12 weeks, allopurinol at a dose of 50 mg/sqm is added (simultaneously reducing the dose of 6MP by 50%) and during the next 12 weeks patients are monitored closely for toxicity and samples for determination of metabolite levels and hematological and liver toxicity are obtained regularly. If, after 4 weeks of allopurinol treatment, the levels of 6-thioguanine are below 200 nmol/mmol hemoglobin, the dose of allopurinol will be increased to 100 mg/sqm. Allopurinol treatment is continued for 12 weeks after which the patients switch to their original maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute lymphoblastic leukemia
* Treatment according to Nordic Society for pediatric hematology/oncology (NOPHO) ALL2008 based protocols
* Age 0-18y at time of initial diagnosis
* TPMT wild type
* Written informed consent

Exclusion Criteria:

* Mature B cell lymphoblastic leukemia
* t(9;22) positive acute lymphoblastic leukemia
* Unknown TPMT status or presence of TPMT mutation (both heterozygous and homozygous)
* Known intolerance to any of the chemotherapeutic drugs in the protocol
* Major organ failure precluding administration of planned chemotherapy
* Severe liver toxicity defined as persistent (≥ two weeks) elevation of either S-bilirubin > 50 μmol/l or S-GPT > 20 x Upper normal limit (UNL) or P-Prothrombin complex > 1.5.
* Reduced kidney function defined as S-creatinine ≥ 1.5 x UNL.
* Lactating female or female of childbearing potential not using adequate contraception.

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
6-thioguanine (6TG) levels in erythrocytes | Up to week 25
  The fraction of patients with 6TG levels over 200 nmol/mmol Hb at week 13 and 25 (ie after 12 weeks standard and allopurinol treatment respectively)

SECONDARY OUTCOMES:
Mean level of 6-thioguanine | Up to week 25
  The mean level of 6TG at week 13 and 25
Mean level of DNA-incorporated thioguanine (DNA-TGN) | Up to week 25
  The mean level of DNA-TGN at week 13 and 25
Mean level of 6-methylmercaptopurine (6MMP) | Up to week 25
  The mean level of 6MMP at week 13 and 25
Mean levels of platelets | Up to week 25
  Comparison of weighted mean of platelets in the treatment phases
Mean levels of hemoglobin | Up to week 25
  Comparison of weighted mean of hemoglobin in the treatment phases
Mean levels of absolute neutrophil count (ANC) | Up to week 25
  Comparison of weighted mean of ANC in the treatment phases
Mean levels of white blood cells (WBC) | Up to week 25
  Comparison of weighted mean of WBC in the treatment phases
Glutamate pyruvate transaminase (GPT) | Up to week 25
  Comparison of weighted means of serum GPT in the treatment phases
Bilirubin | Up to week 25
  Comparison of weighted means of serum bilirubin in the treatment phases
Hypoglycemia | Up to week 25
  Comparison of incidence of hypoglycemia and laboratory measures of metabolic disturbance during the treatment phases
Metabolic disturbance | Up to week 25
  Comparison of incidence of laboratory measures of metabolic disturbance during the treatment phases
Incidence of serious adverse events (SAE) | Up to week 29
  Comparison of the frequency of SAE in the treatment phases
Cumulative dose of 6-mercaptopurine and methotrexate | Up to week 29
  Comparison of the cumulative dose of 6MP and methotrexate and days with treatment interruption in the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Abrahamsson, PhD, MD, Study Chair — Childrens Cancer Center, Queen Silvia Children Hospital, Sahlgrenska Academy, Gothenburg, Sweden; Riita Niinimäki, PhD, MD, Principal Investigator — Dept of Pediatrics and Adolescents, Oulu University Hospital, Box 23, 90029 OYS, Finland
Locations (3):
- Dept of Pediatrics and Adolescents, Oulu University Hospital, Box 23, 90029 OYS, Finland, Oulu, Finland
- Sweden (2):
  - Childrens' Cancer Centre, Queen Silvias Childrens and Adolescents Hospital, Gothenburg
  - Linköping University Hospital, Dept of Pediatrics, Linköping

IPD SHARING:
Plan to Share IPD: No